CLINICAL TRIAL: NCT00701597
Title: Effects of Non-Specific Endothelin-A Receptor Blockade on Ocular Blood Flow in Patients With Glaucoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, Departnebt of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OPHT-020606
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Glaucoma; Blood Flow Velocity
Keywords: ocular blood flow dysregulation, glaucoma, endothelin-1
MeSH Terms: conditions — Glaucoma | interventions — Bosentan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bosentan — Bosentan (Tracleer 125mg Tabletts), peroral, dose: 500mg for 8 days

SUMMARY:
Several lines of evidence suggest now that ocular perfusion abnormalities may contribute to the progression of glaucoma. It has been hypothesised that increased endothelin-1 plasma levels, as seen in patients with glaucoma, may be related to these alterations in ocular blood flow. We could show in recent experiments that administration of ET-1 decreases ocular blood flow, whereas blocking of the ET-A receptors do not affect basal vascular tone in healthy subjects. In the current study we set out to evaluate the effect Bosentan, a non-selective ETA-receptor antagonist in patients with open-angle glaucoma. This should allow us to test the hypothesis that administration of an ET-1 receptor antagonist increases ocular blood flow in patients with glaucoma.

Investigations will be done with a retinal vessel analyzer to determine retinal vessel cross-sectional diameters, with laser Doppler flowmetry and laser Doppler velocimetry to determine subfoveal macular blood flow and optic nerve head blood flow and with laser interferometric measurements to determine fundus pulsation amplitude in the macula. The intraocular pressure will be measured with applanation tonometry. This will be assessed at baseline and in response to peroral application of Bosentan or placebo.

The study objective is therefor, to evaluate the contribution of ET-1 to ocular blood flow dysregulation in patients with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria

* Men and women aged over 18 years
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Inclusion criteria for patients is primary open angle glaucoma defined as pathological optic disc appearance and characteristic visual field loss
* Men and women will be included in equal parts
* Ametropia of less than 6 diopters and anisometropia of less than 2 diopters

Exclusion Criteria (glaucoma patients)

* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Smoking
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Elevated liver enzymes AST and ALT
* Blood donation during the previous 3 weeks
* Ametropy more than 6 dpt
* Systemic treatment with, oral antikoagulation, Glibenclamid or vasoactive drugs
* History of IOP > 30 (untreated)
* Presence of intraocular pathology other than glaucoma
* Advanced visual field defect defined as MD >-10
* Presence of PEX (pseudoexfoliation) glaucoma and pigment glaucoma
* Ophthalmolgical surgery (including argon laser trabeculoplasty (ALT), trabeculectomy, deep sclerectomy) within the last 6 months before the study
* Pregnancy
* Diabetes mellitus

Exclusion criteria (healthy controls)

* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Smoking
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropy more than 6 dpt
* Systemic treatment with oral anticoagulation, Glibenclamid or vasoactive drugs
* Elevated liver enzymes AST and ALT
* Pregnancy
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow (Laser Doppler Flowmetry) Choroidal blood flow(Laser interferometry, Laser Doppler Flowmetry) Retinal blood flow(Laser Doppler velocimetry, Retinal Vessel analyzer) Intraocular pressure (Applanation tonometry) | study 1: ocular blood flow measurements once; study day 2: basline measurements, and after 120min, 180min, 240min after medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjager-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria